CLINICAL TRIAL: NCT03648359
Title: Multiparametric MRI in Men With Prostate Cancer Enrolled in Active Surveillance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Lars Boesen, Primary investigator, MD, PhD, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AS
Record Dates: First submitted 2016-01-19; First posted 2018-08-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate biopsy; Prostate cancer; Magnetic resonance imaging; Neoplasm staging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled AS patients (Other): Patients with prostate cancer enrolled i active surveillance protocol using PSA, digital rectal examination and conventional TRUS-biopsies
  Interventions: Procedure: multiparametric MRI Diagnostics

INTERVENTIONS:
Procedure: multiparametric MRI Diagnostics — Patients with newly diagnosed prostate cancer enrolled in active surveillance following standard protocol including PSA, DRE and TRUS biopsies and intervention with multiparametric MRI + additional biopsies if suspicious lesions are found

SUMMARY:
To investigate whether multiparametric MRI (mp-MRI) in patients with low-risk prostate cancer can improve the selection of patients suitable for Active Surveillance and have a relevance in the ongoing monitoring

DETAILED DESCRIPTION:
Men with localized prostate cancer (PCa) with small tumor burden may be followed on active surveillance (AS) rather than active treatment. AS is an attempt to avoid over-treatment of PCa, which is estimated to be insignificant at the time of diagnosis, and therefore unlikely to affect patient morbidity and mortality. AS include close monitoring with PSA measurement (blood test), digital rectal exploration (DRE) and trans-rectal ultrasound-guided prostate biopsy (TRUS-bx) at regular intervals, so that active treatment can be initiated if the cancer becomes more aggressive. It is crucial that patients undergoing AS are staged correctly, to avoid underestimating more aggressive disease and patients mistakenly are enrolled into AS instead of active treatment.

Previously, a PhD study conducted at Herlev Hospital revealed that multiparametric MRI (mp-MRI) of the prostate can improve the detection and staging of PCa and may add additional information about tumor aggressiveness compared to the traditional methods DRE and TRUS-bx. Mp-MRI at the inclusion of AS may detect missed significant tumors and potential areas of higher aggressiveness than detected by the traditional biopsies. Additional targeted biopsies from these suspicious areas can then be performed with a re-evaluation of the treatment plan, if more advanced disease is identified. Conversely, mp-MRI has a high negative predicted value for significant disease and can be used to rule out significant PCa, reassuring patients and physicians to go on with AS. Mp-MRI has been used at the Urology Department, Herlev Hospital, since 2013 in the diagnosis of PCa and in the evaluation of patients undergoing AS. A retrospective study have show that mp-MRi improve the detection of missed significant PCa.

The main objective of this study is now to prospectively investigate, whether mp-MRI can improve the selection of patients suitable for Active Surveillance and have a relevance in the ongoing monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low risk localized prostate cancer enrolled in active surveillance

Exclusion Criteria:

* Metastatic prostate cancer
* No mp-MRI data present
* Prostate cancer treatment
* Known allergic reaction to Gadolinium-based MRI contrast agent
* Prostate biopsy during the last 21 days
* Impaired renal function with GFR < 30 ml / min
* pacemaker
* Magnetic metal residues in the body
* Claustrophobia
* Psychiatric disorders
* Age under 18 year

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in treatment from active surveillance (observation) to active treatment based on mp-MRI results. | 12 months
  Patients enrolled in active surveillance will progress to active treatment if mp-MRI show previously undetected suspicious areas of significant disease. Significant cancer (measured by Gleason score and cancer core involvement on biopsies) will be confirmed by repeat biopsies of the suspicious areas. The decision to progress to active treatment is based on decision from the treating urologist.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Boesen, MD, PhD, Principal Investigator — Department of Urology, Herlev University Hospital Herleb, Herlev, Denmark, 2730
Locations (1):
- Department of Urology, Herlev University Hospital Herlev, Herlev, Denmark